CLINICAL TRIAL: NCT03381625
Title: A Randomized, Placebo-Controlled, Dose-Escalation Trial to Evaluate the Safety, Clinical Effects, and Systemic Exposure of a Topical Application of BMX-010 in Subjects With Atopic Dermatitis and Plaque Psoriasis
Brief Title: Topical Application of BMX-010 in Subjects With Atopic Dermatitis and Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMimetix JV, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BMX-DERM-01
Record Dates: First submitted 2016-08-18; First posted 2017-12-22 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Psoriasis; Atopic Dermatitis
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMX-010 0.03% (Experimental): 200 subjects will receive BMX-010 0.03% twice daily for 7-28 days applied to psoriasis or atopic dermatitis lesions.
  Interventions: Drug: BMX-010
- Placebo (Placebo Comparator): 100 subjects will receive placebo twice daily for 7-28 days applied to psoriasis or atopic dermatitis lesions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMX-010 — Safety and efficacy of BMX-010 in topical treatment of psoriasis and/or atopic dermatitis.
  Arms: BMX-010 0.03%
Drug: Placebo — Topical administration of placebo in patients with psoriasis and/or atopic dermatitis.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled Phase 2 trial consisting of up to 300 subjects with either psoriasis or atopic dermatitis. In this trial BMX-010 will be topically applied twice daily for up to 28 days.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, multicenter, placebo-controlled study sponsored by BioMimetix JV, LLC (BMX). It is a double-blind parallel cohort study designed to determine the safety and efficacy of BMX-010 (0.03%) relative to Placebo in subjects with atopic dermatitis and psoriasis.

Subjects will be queried regarding adverse events (AEs) and concomitant medication usage.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either atopic dermatitis or psoriasis with mild to moderate lesions involving 1% - 25% of total body surface area
* Candidate for topical treatment of atopic dermatitis or psoriasis
* Negative pregnancy test for females of childbearing potential

Exclusion Criteria:

* Systemic pharmacotherapy or phototherapy for treatment of atopic dermatitis or psoriasis
* Erythrodermic, guttate or generalized pustular psoriasis
* Treatment of systemic retinoids, corticosteroids or immunosuppressive agents within 4 weeks of baseline visit
* Treatment with high potency topical steroids, vitamin D analogs, keratolytics, coal tar, phototherapy, calcineurin inhibitors, or antihistamines within 2 weeks of baseline visit
* UV or Dead Sea therapy within 4 weeks of baseline visit
* Treatment with a biologic agent (monoclonal antibody) within 30 days or 5 times its circulating half-life (whichever is longer) prior to baseline visit
* Atopic dermatitis triggered by environmental allergen or irritant
* Contact dermatitis or drug-induced skin reactions
* Systemic or skin infection requiring antimicrobial therapy
* Systemic chemotherapy or radiotherapy within 4 weeks of baseline visit
* Immunocompromise of any cause
* Pregnancy, lactation or inadequate contraception
* Active drug or alcohol dependence
* Significant acute or chronic medical, neurological or psychiatric illness that would compromise subject's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-07-24 (Actual)

PRIMARY OUTCOMES:
Systemic Adverse Events Caused by BMX-010 on Atopic Dermatitis Lesions | 7-28 days
  Assessment of adverse events occurring following topical administration of BMX-010 to atopic dermatitis lesions
Systemic Adverse Events Caused by BMX-010 on Psoriasis Lesions | 7-28 days
  Assessment of adverse events occurring following topical administration of BMX-010 to psoriasis lesions
Efficacy of BMX-010 against Placebo on Atopic Dermatitis and Psoriasis Lesions | 7-28 days
  Assessment of efficacy

SECONDARY OUTCOMES:
Peak Plasma Concentrations (Cmax) for BMX-010 | 8 days
Area Under the Plasma Concentration Versus Time Curve (AUC) for BMX-010 | 8 days

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Encino Research Center, Encino, California
  - Apex Dermatology, Denver, Colorado
  - Colorado Skin Care, Englewood, Colorado
  - AboutSkin Dermatology & DermSurgery, Greenwood Village, Colorado
  - Ciocca Dermatology, Miami, Florida
  - Dawes Fretzin Dermatology Group, Indianapolis, Indiana
  - Juva Skin & Laser Center, New York, New York
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Dermatology Associates of Nashville, Knoxville, Tennessee
  - Presicion Research Institute, Houston, Texas